CLINICAL TRIAL: NCT07159191
Title: This is a Single-center, Single-arm, Phase II, Prospective Clinical Study Planning to Enroll 30 Patients With Advanced Renal Cell Carcinoma. Eligible Patients, After Signing the Informed Consent Form and Passing the Screening Process, Will Receive Envafolimab + Axitinib Treatment Until Disease Progression or Intolerable Toxicity (Treatment Duration Not Exceeding 24 Months). Clinical Tumor Imaging Assessments Will be Conducted Every 12 Weeks During the Treatment Process According to the RECIST V1.1 Criteria. Safety Will be Assessed Using CTCAE 5.0, With Adverse Events Recorded From Each Treatme
Brief Title: Envafolimab Combined With Axitinib as First-Line Treatment for Patients With Advanced Renal Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-25PJ1755
Record Dates: First submitted 2025-08-18; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Advanced Renal Cell Carcinoma (aRCC)
MeSH Terms: interventions — envafolimab; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Envafolimab + Axitinib (Other)
  Interventions: Drug: Envafolimab Injection, Axitinib Tablets

INTERVENTIONS:
Drug: Envafolimab Injection, Axitinib Tablets — Envafolimab + Axitinib
  * Envafolimab 400 mg, subcutaneous injection, day 1, every 3 weeks;
  * Axitinib 5 mg, orally, twice daily

SUMMARY:
Introduction:

This document explains a clinical research study conducted at Peking Union Medical College Hospital. The study aims to evaluate a new combination treatment - Envafolimab (an immunotherapy) and Axitinib (a targeted therapy) - for patients newly diagnosed with advanced kidney cancer (specifically, clear cell Renal Cell Carcinoma or RCC). This information is designed to help patients, their families, and healthcare providers understand the study's purpose, procedures, potential benefits and risks, and what participation involves.

1. What is the Study About?

   * The Problem: Advanced kidney cancer (RCC) that has spread (metastatic) or cannot be removed by surgery (unresectable) is challenging to treat. While treatments exist, researchers are always looking for more effective and manageable options, especially for patients who haven't had prior systemic (whole-body) anti-cancer therapy.
   * The New Approach: This study combines two types of drugs:

     * Envafolimab: An "immunotherapy" drug given as an injection under the skin (subcutaneous). It works by blocking a protein called PD-L1 on cancer cells or immune cells. Blocking PD-L1 helps the patient's own immune system recognize and attack the cancer cells more effectively.
     * Axitinib: A "targeted therapy" drug taken as a pill twice daily. It works by blocking signals (VEGF receptors) that cancer cells use to grow new blood vessels, essentially starving the tumor of its blood supply.
   * The Goal: To find out if giving Envafolimab and Axitinib together is safe and effective as the first treatment for patients with advanced kidney cancer. Researchers want to see how well the combination shrinks tumors, controls the cancer, and how long patients live without their cancer getting worse, while carefully monitoring side effects.
   * Study Design:

     * Phase II: This is an early stage of testing in patients, focusing mainly on how well the treatment works and its safety profile in a specific group.
     * Single-Arm: All participants in this study will receive the same combination treatment (Envafolimab + Axitinib). There is no separate group receiving a different treatment or placebo for comparison in this particular study.
     * Single-Center: Currently being run at Peking Union Medical College Hospital (but could potentially expand).
     * Participants: Plans to enroll about 30 patients.
     * Treatment Duration: Patients receive treatment as long as it's working (tumor isn't growing) and they can tolerate the side effects, for up to a maximum of 2 years.
2. Key Information for Patients & Families:

   * Who Might Qualify? You may be eligible to participate if you:

     * Are between 18 and 75 years old.
     * Have been diagnosed with advanced clear cell kidney cancer (unresectable or metastatic).
     * Have NOT received any prior systemic anti-cancer treatment (like chemotherapy, immunotherapy, or other targeted therapies) for your advanced kidney cancer.
     * Have tumors that can be measured on scans (CT or MRI).
     * Are relatively active and able to care for yourself (ECOG performance status 0 or 1: meaning you are either fully active or restricted in physically strenuous activity but ambulatory and able to do light work).
     * Have adequate organ function (healthy enough bone marrow, liver, kidneys, heart) as determined by blood tests.
     * Are expected to live at least 6 more months.
     * Understand the study and agree to follow the procedures and attend all visits.
   * Who Would Not Qualify? You would likely not be eligible if you:

     * Have another active cancer besides the kidney cancer being studied.
     * Have had previous systemic treatment for your advanced kidney cancer.
     * Have known severe allergies to similar drugs or components of Envafolimab/Axitinib.
     * Have an active autoimmune disease needing strong medication (like high-dose steroids or immunosuppressants) within the last 2 years. (Hormone replacements like thyroid meds are okay).
     * Are taking high-dose steroids (except inhaled/nasal) or other immune-suppressing drugs shortly before starting.
     * Are using traditional Chinese medicine or immunomodulators within 2 weeks before joining.
     * Have serious uncontrolled heart problems (like recent heart attack, severe heart failure, unstable angina, significant irregular heartbeats).
     * Have uncontrolled fluid build-up needing drainage (like large amounts of ascites or pleural effusion).
     * Are pregnant, breastfeeding, or unwilling to use highly effective contraception during the study and for 6 months after.
     * Have significant psychiatric, substance abuse, or other medical/social issues that the research team believes would interfere with the study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Sign an informed consent form in writing; 2. Age between 18 and 75 years old; 3. Unresectable or metastatic clear cell renal cell carcinoma; 4. No prior systemic anti-tumor treatment; 5. Measurable disease according to RECIST v1.1; 6. ECOG performance status: 0 to 1; 7. Adequate organ and bone marrow function:

  1. Complete blood count: Absolute Neutrophil Count (ANC) ≥ 1.5 × 10^9/L, Platelet (PLT) count ≥ 70 × 10^9/L, Hemoglobin (HGB) ≥ 90 g/L;
  2. Liver function: Total Bilirubin (TBIL) ≤ 1.5 × Upper Limit of Normal Value (ULN); Alanine Aminotransferase (ALT) and Aspartate Transferase (AST) ≤ 3 × ULN; Serum Albumin ≥ 28 g/L; Alkaline Phosphatase (ALP) ≤ 5 × ULN; subjects who meet the above criteria after routine liver protection treatment and have been stable for at least one week after assessment by the researcher can be enrolled;
  3. Renal function: Serum Creatinine (Cr) ≤ 1.5 × ULN, or Creatinine Clearance ≥ 50 mL/min (using the standard Cockcroft-Gault formula);
  4. Coagulation function: International Normalized Ratio (INR) ≤ 1.5 / Prothrombin Time (PT) ≤ 1.5 × ULN, Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 × ULN; if the subject is undergoing anticoagulant therapy, as long as PT and INR are within the range specified for the anticoagulant medication, they are eligible.

  8. Estimated life expectancy ≥ 6 months; 9. Subjects voluntarily participate in this study and have good compliance.

Exclusion Criteria:

* 1. A history of or concurrent with other malignant tumors; 2. Patients who have previously received systemic anti-tumor treatment; 3. Known allergies to macromolecular protein preparations or components of the study medication in the subject's history; 4. Active autoimmune diseases requiring systemic treatment (such as disease-modifying drugs, corticosteroids, or immunosuppressants) have occurred within 2 years prior to the first dose of the study medication. Replacement therapies (such as thyroid hormone, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency, etc.) are not considered systemic treatment; 5. Receiving systemic corticosteroid treatment (excluding nasal, inhalation, or other local routes of administration) or any other form of immunosuppressive therapy within 7 days prior to the first dose of the study medication; Note: The use of physiological doses of corticosteroids (equivalent to ≤50 mg/day of hydrocortisone or equivalent) is permitted; 6. The subject has been using traditional Chinese medicine or other immunomodulators within 2 weeks prior to enrollment; 7. Symptomatic ascites or pleural effusion that cannot be controlled with medication and requires therapeutic puncture or drainage; 8. Uncontrolled cardiac clinical symptoms or diseases, such as:

  1. Heart failure at NYHA class 2 or above;
  2. Unstable angina;
  3. Myocardial infarction within the past year;
  4. Clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention; 9. Known history of abuse of psychiatric drugs, alcoholism, or drug addiction in the subject; 10. Pregnant or nursing women; 11. Men or women of childbearing potential (referring to men or women who have not undergone sterilization surgery, as well as women who have not reached menopause) must use highly effective contraceptive methods (such as oral contraceptives, intrauterine devices, abstinence, or barrier contraception combined with spermicides) during the trial and continue to use contraceptives for 6 months after the last dose; 12. The investigator deems that the subject should be excluded from this study, for example, if the investigator judges that the subject has other factors that may force the study to be terminated prematurely, such as other serious diseases (including psychiatric diseases) requiring concurrent treatment, severe laboratory test abnormalities, or family or social factors that may affect the subject's safety or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-02-20 (Estimated); Study Completion 2027-07-20 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Assessment will be conducted at 6 months, 12 months, 18 months, and 24 months after the intervention begins.

SECONDARY OUTCOMES:
• Disease Control Rate (DCR) | Assessment will be conducted at 6 months, 12 months, 18 months, and 24 months after the intervention begins.
• Progression-Free Survival (PFS) | Assessment will be conducted at 6 months, 12 months, 18 months, and 24 months after the intervention begins.
Overall Survival (OS) | Assessment will be conducted at 6 months, 12 months, 18 months, and 24 months after the intervention begins.
Safety (AE/SAE) | Assessment will be conducted at 6 months, 12 months, 18 months, and 24 months after the intervention begins.
PRO | Assessment will be conducted at 6 months, 12 months, 18 months, and 24 months after the intervention begins.

IPD SHARING:
Plan to Share IPD: No